CLINICAL TRIAL: NCT04244136
Title: Operable Primary Renal Tumors: Pre and Post-operative Volume Evaluation of the Tumor and Rest of the Kidney
Brief Title: Residual Normal Renal Parenchymal and Tumor Volume in Tumor Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohammed ragab abdallah, assistant lecturer in assiut urology hospital,assiut university,Egypt, Assiut University
Other Study IDs: renal tissue volume in tumors
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Renal Cell Carcinoma
Keywords: residual normal renal tissue
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: contrast CT — contrast CT abdomen fir measurement of the volume of expected residual normal renal tissue before surgery

SUMMARY:
1. Calculation of the expected residual renal tissue volume using contrast CT in renal tumor patients and its effect on preoperative decision making
2. Calculating the modulation between the residual normal renal tissue volume measured 6 months post operatively and the preoperative estimated normal renal tissue volume.
3. Assessment of the value of adding residual normal renal tissue volume to the PADUA score in decision making.
4. To reach a suggested cut off value of residual renal tissue that is adequate for a NSS trial

DETAILED DESCRIPTION:
The oncological outcome achieved by NSS is considered equivalent to RN in patients with stage T1 renal tumors and as the benefits of NSS become apparent, the indications and application of NSS continue to expand to involve even higher stages of renal tumors, These trails were successful to achieve nearly a similar oncological outcome, however the functional outcome of the residual renal volume was not calculated because most of these studies depend only on the radiographic stage of the tumor. And it is not logic to expose the patients to the risk of NSS surgery with dissection of a large tumor volume to leave only small residual renal tissue volume that may not have enough benefit. To balance this risk benefit ratio, preoperative assessment of expected residual renal tissue volume can be calculated using contrast CT for all patients with renal masses must be done to reach a cutoff point for the least residual volume of renal tissue that should be left postoperatively to achieve a significant function, and to decide whether to do NSS or to proceed to radical surgery from the start.

The technical skill of the surgeon and the anatomical features of the renal tumor are important factors. The contribution of each factor to treatment choice and outcome are particularly relevant because the physician treatment recommendations are subject to training patterns biases, comfort levels and individual experience also the kidney doesn't follow an anatomical partitioning since designation of independent renal segments based on vascular distributions or collecting duct branching is not possible. Nevertheless, renal anatomy does contain consistent and easily reproducible landmarks which can be used by radiologists and surgeons to describe and quantify pertinent features of renal masses therefore Preoperative Aspects and Dimensions Used for an Anatomical Classification (PADUA) scoring system have emerged for quantifying the anatomical features relevant to surgical decision-making and to predict the risk of surgical and medical perioperative complications in renal tumor patients.

1. Preoperative assessment:

   1. Using contrast CT radiologist will measure the expected residual renal tissue volume ( total renal tissue volume) and PADUA score.
   2. GFR Calculation by Cockcroft-Gault formula.
2. Operative technique:

   NSS will be done whenever possible by open approach, according to PADUA score hot ischemia with clamping of the renal artery will be done in less complicated mass while cold ischemia with cooling of the kidney surface after clamping of both renal artery and vein will be done in more complicated masses, Enculation of the mass will be done whenever possible, excision will be done if needed then closure of renal defect will be done only if necessary.

   Radical nephrectomy will be done only in more complicated cases that are not amenable for NSS by open or laparoscopic approach through early ligation of the renal artery and vein, removal of the kidney outside Gerota's fascia, with or without removal of the ipsilateral adrenal gland, and performance of a complete regional lymphadenectomy whenever possible.
3. Post-operative assessment:

   1. In case of NSS ,immediately post operatively the volume of the mass excised will be measured using graded jar and after 6 months contrast CT for measuring the residual ipsilateral parenchymal renal volume and the volume of the other kidney will be done by the same radiologist who had previously assessed the case (blinded to the preoperative data).
   2. In case of radical nephrectomy, immediately post operatively we will separate the mass from normal renal tissue in the specimen excised then the volume of the mass and the normal renal tissue will be measured using graded jar. After 6 months the volume of the other kidney will be measured by the same radiologist who had previously assessed the case (blinded to the preoperative data)
   3. Residual GFR calculation by GFR Calculation by Cockcroft-Gault formula.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented to oncology outpatient clinic in Assuit urology hospital diagnosed by contrast CT to have renal mass who are surgically fit for radical nephrectomy or NSS surgery.

Exclusion Criteria:

* 1-Patient who diagnosed to have stage T4 renal mass according to TNM staging. 2-CRI patients who cannot perform contrast study. 3-patients with tumors in non-functioning kidney 4-patients with secondary renal tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: renal tumor patients who are fit for renal tumor surgeries
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
estimation of the efficacy of contrast CT IN Calculation of the expected residual normal renal tissue volume before renal tumor surgeries | 3 years
  comparision between preopertive measured volume by CT and post operative measured volume by CT in NSS and by graded gar in radical nephrectomy after isolation of the normal renal tissue in extracted kidney

SECONDARY OUTCOMES:
Assessment of the value of adding residual normal renal tissue volume to the PADUA score in decision making To reach a suggested cut off value of residual renal tissue that is adequate for a NSS trial | 4 years
  study the efficacy of residual normal renal tissue volume in decision making in tumor surgeries and if it have a true rule it what is the cut of value for NSS and can it be added as a fixed measurement to the items of PADUA score

REFERENCES:
- [Background] Long CJ, Canter DJ, Kutikov A, Li T, Simhan J, Smaldone M, Teper E, Viterbo R, Boorjian SA, Chen DY, Greenberg RE, Uzzo RG. Partial nephrectomy for renal masses >/= 7 cm: technical, oncological and functional outcomes. BJU Int. 2012 May;109(10):1450-6. doi: 10.1111/j.1464-410X.2011.10608.x. Epub 2012 Jan 5. PMID 22221502
- [Background] Isotani S, Shimoyama H, Yokota I, Noma Y, Kitamura K, China T, Saito K, Hisasue S, Ide H, Muto S, Yamaguchi R, Ukimura O, Gill IS, Horie S. Novel prediction model of renal function after nephrectomy from automated renal volumetry with preoperative multidetector computed tomography (MDCT). Clin Exp Nephrol. 2015 Oct;19(5):974-81. doi: 10.1007/s10157-015-1082-6. Epub 2015 Jan 25. PMID 25618493
- [Background] Zhang M, Zhao Z, Duan X, Deng T, Cai C, Wu W, Zeng G. Partial versus radical nephrectomy for T1b-2N0M0 renal tumors: A propensity score matching study based on the SEER database. PLoS One. 2018 Feb 28;13(2):e0193530. doi: 10.1371/journal.pone.0193530. eCollection 2018. PMID 29489911
- [Background] Venkatramani V, Swain S, Satyanarayana R, Parekh DJ. Current Status of Nephron-Sparing Surgery (NSS) in the Management of Renal Tumours. Indian J Surg Oncol. 2017 Jun;8(2):150-155. doi: 10.1007/s13193-016-0587-0. Epub 2017 Jan 30. PMID 28546710